CLINICAL TRIAL: NCT04098250
Title: A Multidisciplinary Translational Approach to Investigate the Mechanisms, Predictors, and Prevention of Persistent Post-Traumatic Headache
Brief Title: Multidisciplinary Translational Approach to Investigate Mechanisms Predictors & Prevention of Persistent PTH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Arizona (Other); Translational Genomics Research Institute (Other); Arizona State University (Other); Phoenix VA Health Care System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Amgen (Industry); Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Todd J. Schwedt, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-003200
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Headache
Keywords: headache; post-traumatic headache
MeSH Terms: conditions — Post-Traumatic Headache; Headache | interventions — erenumab

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to erenumab or placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erenumab (Experimental): 140 mg erenumab
  Interventions: Drug: Erenumab
- Placebo (Placebo Comparator): placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Erenumab — a CGRP receptor monoclonal antibody
  Other Names: Aimovig
  Arms: Erenumab
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a United States Department of Defense funded Focused Program study that aims to identify mechanisms and predictors for persistent of post-traumatic headache attributed to mild traumatic brain injury, and identify methods of preventing post-traumatic headache persistence.

The objective of the clinical trial component of the Focused Program is to determine whether intervention with erenumab is an effective treatment for PTH attributed to mTBI.

DETAILED DESCRIPTION:
The human studies component of this Focused Program includes clinical phenotyping, neurophysiology, molecular and genetic biomarker discovery, brain imaging, and a clinical trial.These data will be utilized to characterize post-traumatic headache and build univariate and multivariate predictive models for post-traumatic headache persistence and for the response to post-traumatic headache treatment. These studies are described in more detail within a separate clinicaltrials.gov record.

The clinical trial is a double-blind, randomized, placebo-controlled investigation of erenumab for the treatment of post-traumatic headache. Participants will be randomized when PTH has been present for 35-56 days. Follow-up questionnaires, headache diary data, pain threshold results, and brain imaging data will be collected longitudinally during the clinical trial to assess for changes over time and associations of such changes with post-traumatic headache treatment outcomes. Due to slow enrollment, the study was later changed to open label since the estimated total enrollment would be inadequate for making comparisons between the placebo and erenumab groups.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of acute PTH attributed to mild traumatic injury to the head as defined by the International Classification of Headache Disorders (ICHD-3).
* PTH onset 7-56 days prior to the time of enrollment
* Adults 18-70 years of age
* Willing to be randomized to either of the two clinical trial treatment arms
* Willing to maintain a headache diary
* Willing and able to return for follow-up visits
* 4 or more moderate or severe headache days during the 4-week run-in phase and an increase of at least 2 moderate to severe headache days compared to pre-TBI and at least a 30% increase
* At least 80% compliant with diary keeping during the 4-week run-in phase (i.e., provides data on at least 80% of days)

Exclusion Criteria:

* Chronic headache (i.e., at least 15 headache days/month for more than 3 months) within 12 months prior to the mTBI that led to the current PTH, including PPTH, chronic migraine, medication overuse headache, new daily persistent headache, hemicrania continua, chronic tension-type headache
* Diminished decision-making capacity that in the investigator's opinion would interfere with the person's ability to provide informed consent and complete study procedures
* Started or changed dose of a headache preventive medication within the 3 months prior to screening
* Use of onabotulinumtoxinA in the head, neck or face region within 6 months of screening
* During the 6 months before screening, use of opioids or barbiturates on an average of at least 4 days per month
* Subjects who underwent an intervention or used a device (e.g., nerve blocks, transcranial magnetic stimulation, vagal nerve stimulation, or electrical trigeminal nerve stimulation) for headache within 3 months of screening
* History of major psychiatric disorder such as schizophrenia and bipolar disorder
* History or evidence of any unstable or clinically significant medical condition, that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* History of positive neuroimaging findings that indicate a moderate or severe TBI
* Contraindications to magnetic resonance imaging, including, but not limited to (only an exclusion for patients participating in the brain MRI portion of this research):

  1. Metal implants
  2. Aneurysm clips
  3. Severe claustrophobia
  4. Implanted electronic device
  5. Insulin or infusion pump
  6. Cochlear/otologic/ear implant
  7. Non-removable prosthesis
  8. Implanted shunts/catheters
  9. Certain intrauterine devices
  10. Tattooed makeup
  11. Body piercings that cannot be removed
  12. Metal fragments
  13. Wire sutures or metal staples
* Factors that reduce MR image quality and interpretability (only an exclusion for patients participating in the brain MRI portion of this research):

  1. Dental braces or other non-removable devices (e.g., retainers)
  2. Prior brain surgery
  3. Known brain MRI abnormality that in the investigator's opinion will significantly impact MRI data
* Sensory disorders that in the investigator's opinion might affect perception of cutaneous thermal stimuli (e.g., peripheral neuropathy) (only an exclusion for patients participating in the neurophysiology studies)
* Pregnancy
* Breastfeeding
* History of myocardial infarction, stroke, transient ischemic attack, unstable angina, coronary artery bypass surgery, or other revascularization procedures within 12 months prior to screening.
* Not willing to use a reliable form of contraception (for women of childbearing potential) through 16 weeks after the last dose of erenumab. Acceptable methods of birth control include not having intercourse, hormonal birth control methods, intrauterine devices, surgical contraceptive methods, or two barrier methods (each partner must use a barrier method) with spermicide. A reliable form of contraception must be started prior to or at the time of starting the run-in phase. Not being of childbearing potential is defined as any woman who is post-menopausal by history, defined as:

  1. At least 55 years of age with cessation of menses for 12 or more months; OR
  2. Younger than 55 years of age but no spontaneous menses for at least 2 years; OR
  3. Younger than 55 years of age and spontaneous menses within the past 1 year, but currently amenorrheic (e.g., spontaneous or secondary to hysterectomy), AND with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels at least 40 IU/L) or postmenopausal estradiol level (less than 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved; OR
  4. Underwent bilateral oophorectomy; OR
  5. Underwent hysterectomy; OR
  6. Underwent bilateral salpingectomy.
* Currently or within 90 days prior to screening: received treatment in another drug study or an investigational device study
* Has previously received any CGRP ligand or receptor targeted monoclonal antibody

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schwedt, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mayo Clinic Arizona.
Pre-assignment Details: All subjects who participated in the study took part in the trial prior to the study team changing it to an open label study. No participants were recruited or enrolled after the study was changed to open label.
Period: Overall Study
Arm/Group | Erenumab | Placebo
Started | 2 | 4
Completed | 1 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erenumab | Placebo | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (10.2) | 42.3 (26.0) | 43.9 (20.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Days Experiencing Moderate-to-Severe Headaches
Description: The number of days where subjects experienced moderate-to-severe headaches. This was measured at baseline, 9, 10, 11 and 12 weeks after administration of first dose of erenumab 140 mg or placebo. The change from baseline to week 12 is reported.
Time Frame: Baseline, 9, 10, 11 and 12 Weeks, change from baseline to week 12 reported
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 2 | 3
Days | -8 (2.8) | -0.33 (6.0)

2. Secondary Outcome: Responder Rate
Description: The number of patients with at least a 50% reduction in days where they experienced a headache. This was measured at baseline, 9, 10, 11 and 12 weeks after administration of first dose of erenumab 140 mg or placebo. The change from baseline to week 12 is reported.
Time Frame: Baseline, 9, 10, 11 and 12 Weeks, change from baseline to week 12 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 1 | 1

3. Secondary Outcome: Chronic Headache
Description: The number of patients with a chronic headache, defined as reporting a headache for at least 15 days. This was measured at baseline, 9, 10, 11 and 12 weeks after administration of first dose of erenumab 140 mg or placebo. The change from baseline to week 12 is reported.
Time Frame: Baseline, 9, 10, 11 and 12 Weeks, change from baseline to week 12 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 1 | 1

4. Secondary Outcome: Change in the Headache Impact Test (HIT-6)
Description: The Headache Impact Test (HIT-6) measures the impact of headaches on a person's daily life. It assesses the frequency and severity of headaches, their functional limitations and the impact on daily activities such as work, education and social interactions. The HIT-6 test has 6 questions. Each of the six questions receives a score from 6-13. The final HIT-6 score can range from 36 to 78. A higher score indicates more disability due to headache. This was measured at baseline, 9, 10, 11 and 12 weeks after administration of first dose of erenumab 140 mg or placebo. The change from baseline to week 12 is reported.
Time Frame: Baseline, 9, 10, 11 and 12 Weeks, change from baseline to week 12 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 2 | 4
score on a scale | -7 (1.4) | -1.3 (14.4)

5. Secondary Outcome: Change in the Number of Days Where Acute Treatment Was Administered to Relieve a Headache
Description: The change in the number of days where subjects underwent acute treatment to relieve a headache. Treatment days were days in which subjects took analgesic, triptan, or ergotamine containing medication, or they underwent device neuromodulation [e.g. vagal or trigeminal nerve electrical stimulation or single pulse transcranial magnetic stimulation]. This was measured at baseline,9, 10, 11 and 12 weeks after administration of first dose of erenumab 140mg or placebo. The change from baseline to 12 weeks is reported.
Time Frame: Baseline, 9, 10, 11 and 12 Weeks, change from baseline to week 12 reported
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 2 | 3
Days | -7.5 (4.9) | -2.7 (4.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the first dose of investigational product through the end of the safety follow up visit, approximately 12 weeks.
Arm/Group | Erenumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erenumab (N=2) | Placebo (N=4)
Pain at injection site/bruising at injection site (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2)
COVID (Infections and infestations) | 1 (1) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia/Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Eyelid Twitching (Eye disorders) | 0 (0) | 1 (1)
Facial Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Dizziness/Increased Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT04098250/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT04098250/ICF_002.pdf